CLINICAL TRIAL: NCT03714932
Title: Accuracy of Arch Analysis in Mixed Dentition Using Digital Study Models Versus the Plaster Models Using Tanaka and Johnston Prediction Equation:
Brief Title: Accuracy of Arch Analysis in Mixed Dentition Using Digital Models Versus Plaster Ones.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Tag El Deen, Master student in Cairo university (principle Invistigator), Cairo University
Other Study IDs: CEBD-CU-2018-09-36
Record Dates: First submitted 2018-10-01; First posted 2018-10-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2019-10

CONDITIONS: Dental Malocclusion
Keywords: Arch analysis, Mixed dentition,Tanaka & Johnston
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3shape ortho analyzer software — Arch analysis , manual analysis , digital analysis , Mixed dentition , Tanaka and Johnston

SUMMARY:
Accuracy of arch analysis in mixed dentition using digital study models versus the plaster models using Tanaka and Johnston prediction equation:

DETAILED DESCRIPTION:
Space analysis is traditionally performed by diagnostic measurements that have been obtained from plaster dental casts through measurements which might be influenced by subjective interpretation and bias when constructed.

*So another method of diagnostically measuring study models was introduced (Digital software). This system creates digital images of dental casts with software. From the digitized models, various analyses and routine measurements could be done that might accelerate and solve many problems and difficulties associated with storage, retrieval, reproduction, communication, and breakage of conventional plaster casts.

* Taking an impressions for a mixed dentition aged children.
* Perform a measurements using Tanaka and Johnston equation for an arch analysis using a caliper and 3Shape ortho-analyzer software.
* Casts will be scanned using the 3D scanner then by using the 3shape software measurements will be held according to Tanaka and Johnstopn prediction equation.

ELIGIBILITY:
Inclusion Criteria:

* Aged range from 6-10.
* patients medically free from any syndromes that could affect the normal eruption.
* Normal radiographical findings in teeth eruption.
* Erupted lower incisors.

Exclusion Criteria:

* Extracted lower 1st permanent molar.
* congenital missing of incisors.
* Badly decayed permanent incisors or 1st molar that could compromise the measurements.
* Any sensitivity to any of the impression materials.

Ages: 6 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Children aged six to Ten years.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
accuracy of digital models in arch analysis. | 6 months
  using digital models through software(3shape ortho analyzer) to evaluate it's accuracy in arch analysis through prediction equation(Tanaka and Johnston equations)versus plaster models by using manual caliper.

CONTACTS AND LOCATIONS:
Overall Officials: sara Mohamed Tag El Deen, Master, Study Director — Cairo University
Locations (1):
- sara Mohamed, Cairo, Egypt